CLINICAL TRIAL: NCT05501262
Title: Comparative Effectiveness of Cryoablation Using the ICE-Seed Cryoablation Needle With Steroid and Lidocaine Versus Steroid and Lidocaine Alone for Treatment of Morton's Neuroma
Brief Title: Comparative Effectiveness of Cryoablation Versus Steroid and Lidocaine Alone for Treatment of Morton's Neuroma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Boston Scientific Corporation (Industry); Society of Interventional Radiology Foundation (Other)
Responsible Party: Principal Investigator, Claire Kaufman, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00024090
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Morton Neuroma
MeSH Terms: conditions — Morton Neuroma | interventions — Cryosurgery; Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Steroid and lidocaine injection
  Interventions: Procedure: Nerve block
- Study (Experimental): Steroid and lidocaine injection with cryoablation
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Image (ultrasound and fluoroscopic guided) cryoablation will be performed of the Morton's neuroma after nerve block.
  Arms: Study
Procedure: Nerve block — Ultrasound and fluoroscopic guided nerve block.
  Arms: Standard of Care

SUMMARY:
Morton's neuroma is a benign thickening involving the plantar interdigital nerve, most common in middle aged women. Morton's neuroma is one of the most frequent diagnoses seen in the investigators podiatry clinic and is difficult to treat. These lesions cause a burning or shooting pain that can radiate to the toes, or an aching pain in the ball of the foot. The pain is exacerbated with activity and certain footwear greatly limits activity in the involved patient population. Morton's neuroma is first treated conservatively with orthotics. Patients may require further interventions such as steroid injections. The literature reports only a 30% long term resolution of pain with the steroid. Surgical resection has a reported 51-85% success rate with 14-21% rate of complication; recurrent pain, numbness/loss of sensation, and subsequent stump neuromas.

Cryoablation is well known to be efficacious for neuropathic pain and has recently been shown in two small studies to be safe and efficacious for treatment of Morton's neuroma. The investigators study will compare outcomes of cryoablation to corticosteroid injection in short- and long-term for treatment of Morton's neuroma that have failed conservative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to consent and complete questionnaires
* Failure of a four-week trial of conservative therapy (includes orthotics, appropriate footwear, and/or metatarsal pads)
* X-ray and ultrasound excluding other pathology and confirming the presence and location of a Morton's neuroma

Exclusion Criteria:

* Inability to follow-up or to comply with the follow-up protocol
* Contraindication to cryoablation and/or lidocaine/steroid injection
* Other pathology which could account for symptoms identified on imaging studies
* Unwillingness to be randomized

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life | 1 year post procedure
  Will be evaluated using the SF-36 Quality of Life Survey
Réponse in pain | 1 year post procedure
  Will be evaluated using the visual analog scale with 0 as no pain and 10 as the word pain imaginable
Changes to function | 1 year post procedure
  Changes to the modified American Orthopedic Foot and Ankle Society Hallux Metatarsophalangeal--Interphalangeal Scale, higher score is less symptomatic
Changes pain and function due to neuroma | 1 year post procedure
  Changes in Neuroma Scale, higher score is less symptomatic
Incidence of Treatment - Emergent Adverse Events | 1 year post procedure
  Monitoring for safety of the treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Claire Kaufman, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be shared with other researchers via a secure web based portal.